CLINICAL TRIAL: NCT01793493
Title: Effects of Cognitive Stimulation in Elderly Individuals at Risk to Develop Dementia: a Randomized Controlled Trial (Allena-Mente).
Brief Title: Cognitive Stimulation in Elderly Individuals at Risk to Develop Dementia (Allena-Mente).
Acronym: Allena-Mente
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Golgi Cenci (Other)
Collaborators: Alzheimer Federation Italy (Other); Camillo Golgi Geriatric Institute (Other); University of Pavia (Other); Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Principal Investigator, Antonio Guaita, MD, MD, Fondazione Golgi Cenci
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment; Healthy Subjects With Family History for Dementia
Keywords: Mild Cognitive Impairment; Cognitive Stimulation; Aging; Elderly; Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive stimulation (Experimental)
  Interventions: Other: Cognitive stimulation
- Sanitary education (Active Comparator)
  Interventions: Other: Sanitary education

INTERVENTIONS:
Other: Cognitive stimulation — Participants are pooled in small groups (6-8 individuals). Each group participates to ten twice weekly meetings. Each CS session is run by one trained operator. One observer participates to the sessions to guarantee homogeneity between different operators. Exercises are structured with an increasing cognitive complexity and are tailored to the characteristics of the group.
  Meetings (each lasting about 2 hours) have a common structure:
  * body awakening (10 minutes)
  * cognitive stimulation (1 hour and a half) scheduled as follow:
    * temporospatial orientation
    * attentional abilities
    * one of the following cognitive areas: language, executive functions, verbal and visual memory (encoding, consolidation, retrieval)
  Arms: Cognitive stimulation
Other: Sanitary education — Participants attend two weekly meetings (for a total of 3 hours) focused on lifestyle education and brain functioning.
  Arms: Sanitary education

SUMMARY:
The Allena-Mente study is a randomized, controlled, single-blind trial assessing the efficacy of cognitive stimulation (CS) compared to an active control group, participating to sanitary education lessons (AC). This non-pharmacological intervention is delivered to Mild Cognitive Impairment (MCI) and cognitively healthy individuals with first-degree relative with dementia (NDFAM).

DETAILED DESCRIPTION:
The experimental protocol was set up with a pilot study on healthy elderly individuals. Data from this pilot study will be excluded from the statistical analysis.

Sample size: a priori power analysis was performed to evaluate the sample size required for the study. MCI and NDFAM were considered separately for sample size calculation. For power calculation a two-tailed test was used and a significance level (α) and test power (1-β) were set at 0.05 and 0.8/0.9, respectively.

Randomization: The individuals belonging to MCI and NDFAM subgroup were randomly assigned to CS or AC group. The randomization was performed by a statistician blind to participants characteristics using the Random Allocation Software. Allocation ratio was set at 1:1, stratification was performed for birth cohort (≤1937 and ≥1938), education level (years of education ≤5 years and >5 years).

Participants provided written informed consent before study participation.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis for mild cognitive impairment (MCI) according to Petersen's criteria;
* Cognitively healthy elderly individuals, having at least one first-degree relative affected by dementia (Alzheimer's Disease, pre-senile and senile dementia, vascular dementia) (NDFAM).

Exclusion Criteria:

* (Major physical illness) Compromission of motor performance of lower and upper limbs
* Medical conditions leading to clinical instability;
* Therapies that reduce cognitive and communicative abilities and consciousness;
* Perceptual disorders (sight, hearing)
* Language disorders
* Education level lower than 3 years
* Psychiatric and behavioral disorders
* Addiction to drugs or alcohol

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Long-term change from Baseline in Mini Mental State Examination (MMSE) | baseline and up to 4 years
  Mini Mental State examination (MMSE) is a brief test of mental status and cognitive function, commonly used in clinical research to screen global cognitive functioning.

SECONDARY OUTCOMES:
Change from Baseline in Mini Mental State Examination at 2-weeks after the intervention | baseline, two-weeks after the intervention
  MMSE is a brief test of mental status and cognitive function, commonly used in clinical research to screen global cognitive functioning.
Change from Baseline in Montreal Cognitive Assessment (MoCA) at 2-weeks after the intervention | baseline, two-weeks after the intervention
  MoCA is a brief cognitive screening tool with a high sensitivity and specificity for detecting MCI in individuals performing in the normal range on the MMSE (avoiding ceiling effect).
Change from Baseline in Corsi test at 2-weeks after the intervention | baseline, two-weeks after the intervention
  Corsi test evaluates visual-spatial short-term memory. We used this test to implement non-verbal memory in our neuropsychological test battery
Change from Baseline in Walking While Talking Dual Task at 2-weeks after the intervention | baseline, two-weeks after the intervention
  Walking speed measures the ability to perform a dual action task. Single task: participants walk back and forth along an indicated distance of 5 meters with no pausing.
  Dual task: participants perform the same movement as in the single task while listing personal names in a loud voice (female names for men and male names for women) The span between time needed to perform the dual and the single task is registered.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Guaita, MD, Study Director — GolgiCenci Foundation
Locations (1):
- Golgi Cenci Foundation, Abbiategrasso, Milan, Italy

REFERENCES:
- [Background] Polito L, Abbondanza S, Vaccaro R, Valle E, Davin A, Degrate A, Villani S, Guaita A. Cognitive stimulation in cognitively impaired individuals and cognitively healthy individuals with a family history of dementia: short-term results from the "Allena-Mente" randomized controlled trial. Int J Geriatr Psychiatry. 2015 Jun;30(6):631-8. doi: 10.1002/gps.4194. Epub 2014 Sep 3. PMID 25187003
- See also: official web site of the organization responsible for the study — http://www.golgicenci.it
- See also: official website of the caregivers organization, partner in the sponsorship of the research — http://www.alzheimer.it